CLINICAL TRIAL: NCT00512668
Title: Phase Ib Study of Limited Androgen Ablation and Two Dose Levels of Temsirolimus (NSC#683864) in Patients With Prostate Cancer Who Have a Biochemical Relapse After Prostatectomy and/or Radiotherapy
Brief Title: Hormone Therapy and Temsirolimus in Treating Patients With Relapsed Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03098; 2007-0025
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Goserelin; bicalutamide; nilutamide; Flutamide; temsirolimus; Sirolimus

ARMS (1):
- Treatment (hormone therapy, temsirolimus) (Experimental): Patients receive combined androgen ablation therapy comprising a luteinizing hormone-releasing hormone analogue (i.e., leuprolide acetate intramuscularly once monthly or goserelin subcutaneously every 3 months) and an oral anti-androgen drug (i.e., bicalutamide or nilutamide once daily or flutamide 3 times daily) on days 1-90.* Beginning on day 60 of hormonal therapy, patients receive temsirolimus IV over 30 minutes once weekly. Treatment with temsirolimus continues for up to 36 weeks in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients may receive no more than 3 months of hormonal therapy, including therapy initiated within 2 months of study entry.
  Interventions: Drug: leuprolide acetate; Drug: goserelin acetate; Drug: bicalutamide; Drug: nilutamide; Drug: flutamide; Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: leuprolide acetate — Given intramuscularly
  Other Names: Enantone; LEUP; Lupron; Lupron Depot
Drug: goserelin acetate — Given subcutaneously
  Other Names: ICI-118630; ZDX; Zoladex
Drug: bicalutamide — Given PO
  Other Names: Casodex; CDX
Drug: nilutamide — Given PO
  Other Names: ANAN; Anandron; Nilandron
Drug: flutamide — Given PO
  Other Names: Eulexin; Eulexine; FLUT; Sch 13521
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given together with hormone therapy in treating patients with relapsed prostate cancer. Androgens can cause the growth of prostate cancer cells. Hormone therapy may fight prostate cancer by lowering the amount of androgens the body makes. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving hormone therapy together with temsirolimus may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize safety and drug-related adverse events of two doses (15 and 25 mg) of intravenous weekly temsirolimus combined with short term complete androgen ablation and to select a favorable and tolerable dose for prostate cancer patients who experience biochemical failure after prostatectomy and/or radiation therapy.

SECONDARY OBJECTIVES:

I. To archive tissue and blood components for future study of molecular markers of response and disease progression.

II. To evaluate the effects of 2 dose levels of temsirolimus on changes in the phosphorylation state of proteins in the mTOR pathway using western blots on peripheral blood mononuclear cells (PBMCs).

OUTLINE:

Patients receive combined androgen ablation therapy comprising a luteinizing hormone-releasing hormone analogue (i.e., leuprolide acetate intramuscularly once monthly or goserelin subcutaneously every 3 months) and an oral anti-androgen drug (i.e., bicalutamide or nilutamide once daily or flutamide 3 times daily) on days 1-90.* Beginning on day 60 of hormonal therapy, patients receive temsirolimus IV over 30 minutes once weekly. Treatment with temsirolimus continues for up to 36 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may receive no more than 3 months of hormonal therapy, including therapy initiated within 2 months of study entry.

After completion of study therapy, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must also have signed an authorization for the release of their protected health information
* Patients must have histologically confirmed adenocarcinoma of the prostate recurring after local therapy (radical prostatectomy and/or radiation therapy) as evidenced by rising serum PSA
* Prostate-Specific Antigen (PSA) Doubling Time (PSADT) =< 12 months after local therapy (prostatectomy and/or definitive radiation) as determined by linear regression of all available PSA values within 6 months of initiation of androgen ablation (for patients who underwent prostatectomy, at least one PSA measurement of >= 1.0 ng/mL; for patients who underwent radiation, at least one PSA measurement of >= 3.0 ng/mL and >= 150% postradiation nadir)
* No evidence of metastasis as determined by bone scan or computed tomography (CT) scan
* Initiation of Androgen Ablation of less than 8 weeks' duration prior to study entry is permitted
* Leukocytes ≥ 3,000/mcl
* Absolute neutrophil count ≥ 1,000/mcl
* Hemoglobin ≥ 8.0g/dl

  * Eligibility level for hemoglobin may be reached by transfusion
* Platelet count >= 100,000/μL
* Total bilirubin ≤1.5 X laboratory ULN
* AST and/or ALT ≤ 3 X laboratory ULN
* Creatinine ≤ 1.5 X laboratory ULN OR calculated creatinine clearance ≥ 60 ml/min/1.73 m^2 for patients w/creatinine levels above the laboratory ULN
* Serum cholesterol level < 350 mg/dl
* Triglyceride level < 300mg/dl
* ECOG performance status 0, 1 or 2
* The effects of Temsirolimus on the developing human fetus are unknown; for this reason men must agree to use contraception from the time of study enrollment continuing for the duration of study participation
* Patients must be registered in the MDACC institutional database prior to treatment with study drug
* PSA < 40 ng/ml

Exclusion Criteria:

* Patients with histologic variants other than adenocarcinoma in the primary tumor
* Patients may not be receiving any other investigational agents
* Patients may not be receiving concomitant immunotherapy or immunosuppressive therapy
* Patients may not have received prior systemic treatment for prostate cancer (other than no more than 3 months of prior treatment with androgen ablation in neoadjuvant and/or adjuvant setting and at least a year must have elapsed since last administration) unless initiation of Androgen Ablation of less than 8 weeks' duration prior to study entry is permitted
* Patient with uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring parenteral therapy on day 1 of protocol treatment, symptomatic congestive heart failure resulting in a resting O2 saturation of < 92% on room air, unstable angina pectoris, myocardial infarction within the previous 6 months, or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia, known pulmonary hypertension or pneumonitis
* Patients in a severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV) due to possible pharmacokinetic interactions with HAART therapy
* Patients diagnosed with acute or chronic hepatitis B or C
* Patients using immunosuppressive agents, including intravenous corticosteroids, within 3 weeks of study entry
* Patients must not have a history of any other cancer (except nonmelanoma skin cancer), unless in complete remission and off of all therapy for that disease for a minimum of 3 years

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety, in terms of drug-related adverse events of two doses of temsirolimus following androgen ablation | 180 days
Favorable and tolerable dose for prostate cancer patients who experience biochemical failure after prostatectomy and/or radiation therapy | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States